CLINICAL TRIAL: NCT03282383
Title: Shanghai Changhai Hospital,Second Military Medical University
Brief Title: Identification of Biomarkers for Severe Pneumonia
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, changhai hospital, Changhai Hospital
Other Study IDs: Severe pneumonia biomarkers
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Biomarkers
Keywords: biomarkers pneumonia severity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the potential serum biomarkers with regard to the severity of pneumonia, and to further evaluate the prognostic value of these markers.

DETAILED DESCRIPTION:
First, we will collect serum samples from patients with pneumonia. Then we will identify biomarkers differentially expressed between non-severe pneumonia and severe pneumonia. We will further evaluate the prognostic value of these markers for pneumonia.

ELIGIBILITY:
Inclusion Criteria:

- under 18 years old

Exclusion Criteria:

* over 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: collection the blood from 600 patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
microRNA | 3 years
  the all of microRNA of blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Kong, MD, Principal Investigator — Changhai Hospital